CLINICAL TRIAL: NCT06699615
Title: Survey of Medical Oncologists to Assess Trustworthiness of Various Approaches to AI Explainability for Prognostic Models
Brief Title: Assessing Perceptions of ML Explanations by Medical Oncologists
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 29524; 857324 (Registry Identifier: UPENN IRB)
Record Dates: First submitted 2024-11-19; First posted 2024-11-21 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-01

CONDITIONS: Oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Consented participants will complete a one time de-identified Qualtrics survey.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- One time de-identified Qualtrics Survey (Other)
  Interventions: Other: Once time de-identified Qualtrics survey

INTERVENTIONS:
Other: Once time de-identified Qualtrics survey — Once time de-identified Qualtrics survey

SUMMARY:
The objective of this proposal is to conduct a vignette-based survey among practicing oncology clinicians who treat non-small cell lung cancer to assess the trustworthiness of explainable predictions from a neurosymbolic AI vs. State-of-the-art post-hoc explanatory algorithms, using simulated patient data.

ELIGIBILITY:
Inclusion Criteria "Medical oncologist" or "Hematologist/Oncologist" designation at Penn Treats lung cancer

Exclusion Criteria:

Non-medical oncologists No email address or physical address listed Does not treat lung cancer

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Determine whether neurosymbolic AI explainability methods improve the trustworthiness of explanations from a prognostic model, relative to post-hoc explainers. | 3 months
  Oncologist will be invited to complete a vignette-based survey

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States